CLINICAL TRIAL: NCT04315649
Title: Effect of 3D Movie Viewing on Stereopsis in Strabismus and / or Anisometropic Amblyops
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Politècnica de Catalunya (Other)
Collaborators: Hospital Mutua de Terrassa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PhDLAJE2
Record Dates: First submitted 2020-03-16; First posted 2020-03-19 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Amblyopia; Anisometropic Amblyopia; Strabismic Amblyopia
Keywords: 3D movies; Amblyopia treatment
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 3D movie (Experimental): 3D movie viewing
  Interventions: Other: 3D movie viewing

INTERVENTIONS:
Other: 3D movie viewing — 3D movie viewing

SUMMARY:
This study evaluates the effect of 3D movie viewing on stereopsis recovery in anisometropic and / or strabismus amblyopia and the satisfaction with the intervention.

DETAILED DESCRIPTION:
Amblyopia is a visual neurodevelopmental disorder associated, more frequently, with the presence of strabismus and anisometropia. It is clinically most important visual condition in childhood because, apart from refractive error, it is the most frequent cause of vision loss in children. It is a reversible condition that affects up to 5% of the population, and that is the result of an abnormal visual experience during the most sensitive period of visual development. Although amblyopia is expressed in the clinical practice as a reduction in visual acuity, it is also characterized by an altered stereoscopy. Generally, treatments for amblyopia focus on the recovery of visual acuity, and there are no treatments that focus mainly on the recovery of the altered stereopsis, so present and with an important functional impact.

The aim of this study reviewing, analyzing and, if applicable, updating the current treatment model for amblyopia. On the one hand, to evaluate the effectiveness of viewing a 3D movie in the improvement of stereoacuity and the deviation, as well as visual acuity and sensitivity to contrast. Also, the correlation between them. On the other hand, to assess quantitatively the degree of satisfaction and acceptance of the participants and their families towards the intervention.

A quasi-experimental study will be performed, without a control group, pre- and post- intervention in which subjects with refractive and / or strabismus amblyopia, that have been subjected to traditional treatment for amblyopia, will be selected. Variables of stereopsis, latent or manifest deviation, visual acuity and sensitivity to the contrast will evaluate previously and after the intervention.

The sample will include subjects between 5 to 12 years old with a diagnosis of refractive and / or strabismic amblyopia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of refractive and / or strabismus amblyopia at some point in life
* History of amblyopia treatment completed at least 6 months before the intervention
* Deviation angle equal to or less than 10 Dp
* Absence of associated ophthalmological pathology.

Exclusion Criteria:

* Ongoing amblyopia treatment;
* Non-comitant and/or large constant strabismus (>10 prism diopters)
* Any ocular pathological condition or nystagmus.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline Stereopsis, immediately after intervention and at 3 months studying the effect of viewing a 3D movie on visual function. | Baseline, immediately after intervention and 3 months
  Stereopsis (ST in logMAR) will be evaluated by a TNO test.
Change from baseline latent or manifest deviation at 6m, immediately after intervention and 3 months studying the effect of viewing a 3D movie in the visual function. | Baseline, immediately after intervention and 3 months
  Latent o manifest deviation will be evaluated at 6 m and will be measured by prisms.
Change from baseline latent or manifest deviation at 40cm, after intervention at and 3 months studying the effect of viewing a 3D movie in the visual function. | Baseline, immediately after intervention and 3 months
  Latent o manifest deviation will be evaluated at 40cm and will be measured by prisms.

SECONDARY OUTCOMES:
Satisfaction assessed by an ordinal questionnaire designed based on the Treatment Satisfaction Questionnaire for Medication (TSQM). | Immediately after intervention
  Satisfaction assessed by an ordinal questionnaire (1 to 5, as 1 the lowest satisfaction and 5 the highest satisfaction), based on the TSQM (Treatment Satisfaction Questionnaire for Medication) version 1.4 to provide data regarding the degree of satisfaction and sensation of parents and children in relation to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Asensio Jurado, MsC, Principal Investigator — Universitat Politècnica de Catalunya; Marc Argilés Sans, PhD, Study Director — Universitat Politècnica de Catalunya; Lluïsa Quevedo i Junyent, PhD, Study Director — Universitat Politècnica de Catalunya
Locations (1):
- Laura Asensio Jurado, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bridgeman B. Restoring adult stereopsis: a vision researcher's personal experience. Optom Vis Sci. 2014 Jun;91(6):e135-9. doi: 10.1097/OPX.0000000000000272. PMID 24811849
- [Background] Levi DM, Knill DC, Bavelier D. Stereopsis and amblyopia: A mini-review. Vision Res. 2015 Sep;114:17-30. doi: 10.1016/j.visres.2015.01.002. Epub 2015 Jan 29. PMID 25637854
- [Background] Li RW, Tran KD, Bui JK, Antonucci MM, Ngo CV, Levi DM. Improving Adult Amblyopic Vision with Stereoscopic 3-Dimensional Video Games. Ophthalmology. 2018 Oct;125(10):1660-1662. doi: 10.1016/j.ophtha.2018.04.025. Epub 2018 May 18. No abstract available. PMID 29779684
- [Background] Birch EE, Jost RM, De La Cruz A, Kelly KR, Beauchamp CL, Dao L, Stager D Jr, Leffler JN. Binocular amblyopia treatment with contrast-rebalanced movies. J AAPOS. 2019 Jun;23(3):160.e1-160.e5. doi: 10.1016/j.jaapos.2019.02.007. Epub 2019 May 16. PMID 31103562
- [Background] Bossi M, Tailor VK, Anderson EJ, Bex PJ, Greenwood JA, Dahlmann-Noor A, Dakin SC. Binocular Therapy for Childhood Amblyopia Improves Vision Without Breaking Interocular Suppression. Invest Ophthalmol Vis Sci. 2017 Jun 1;58(7):3031-3043. doi: 10.1167/iovs.16-20913. PMID 28614556